CLINICAL TRIAL: NCT06664892
Title: Ultrahypofractionated Whole Breast Radiation Following Breast Conserving Surgery and Chemotherapy in Patients > 60 Years of Age With Clinically Low-Risk, Node-Negative Breast Cancer Who Have Received Prior Chemotherapy
Brief Title: Ultrahypofractionated Whole Breast Radiation Following Chemotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MHCI 24-01
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Radiation: Ultra-hypofractionated radiation

INTERVENTIONS:
Radiation: Ultra-hypofractionated radiation — RT, delivered via external beam, 5.2 Gy per fraction for 5 fractions following BCS and neoadjuvant or adjuvant chemotherapy. Specific adjuvant/neoadjuvant therapies are at the discretion of the treating Medical Oncologist.

SUMMARY:
This is a single institution, non-randomized, non-inferiority study comparing prospectively collected data for acute and late effects on the breast associated with ultrahypofractionated whole breast radiation (WBI) following breast conserving surgery (BCS) and chemotherapy to historical controls for breast cancer (BC) patients who receive hypofractionated RT following BCS and chemotherapy.

DETAILED DESCRIPTION:
Standard treatment approaches for patients with localized BC includes BCS followed WBI [1], which has demonstrated equivalent local control and survival when compared to mastectomy [2,3]. Although conventionally fractionated radiotherapy (RT) (50 Gy 2 Gy per fraction) administered in 25 fractions in 5 weeks was historically used, moderate hypofractionation RT trials utilizing shorter treatment times and higher doses per session have resulted in favorable outcomes [4,5,6]. In addition, increased local control and reduced toxicity rates observed in moderate hypofractionation RT trials [5,6] have resulted in studies evaluating the use of ultrahypofractionated breast RT which further shorten the treatment time. The results of the FAST-Forward RT trial have shown that adjuvant RT using 26 Gy/5.2 Gy per fraction, over 5 fractions administered in 1 week, was not inferior to the standard 40.05 Gy/15 fx/3 weeks for local tumor control and is equally safe in terms of effects on normal tissue [7]. Side effects associated with RT can be more pronounced in patients when RT is combined with surgery and/or chemotherapy [9]. There are abundant data describing the safety of combining conventionally fractionated RT following chemotherapy. Similarly, there are several trials which have reported outcomes of patients who have received hypofractionated RT, including subsets of patients who also received chemotherapy demonstrating similar acute and late toxicity profiles compared to standard fractionation regimens [10, 11, 12, 13]. Although the FAST-Forward trial included patients who received neoadjuvant and adjuvant chemotherapy and estimates of 5-year cumulative incidence of any moderate or marked clinician-assessed normal tissue effects in the breast or chest wall were reported to be similar for 40 Gy 15 fraction hypofractionated vs the 26 Gy 5 fraction ultrahypofractionated RT regimen (26·8% v 28·5%, respectively), the study was not designed to detect differences for those who had received prior chemotherapy compared to those who did not [7]. Retrospective subgroup analysis did not identify differences in adverse effects related to prior chemotherapy, however confidence intervals overlapped, and the power for these retrospective subgroup analyses was low [19]. Hence, there is limited data evaluating the toxicity of ultrahypofractionated adjuvant breast RT in patients who have received prior chemotherapy. This study is designed to evaluate the acute and late effects on the breast of ultrahypofractionated WBI using the FAST-forward regimen (26 Gy, 5.2 Gy per fraction delivered in 1 week) in patients > 60 years of age with pathologically or clinically node-negative early-stage BC who undergo BCS and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged at least 60 years with invasive BC (T1-3) with clinically or pathologically negative axillary nodes following BCS who have a high-risk Mammaprint or Oncotype testing and receive chemotherapy. (If no axillary surgery planned, patients must have pre-operative negative axillary ultrasound)
2. Invasive ductal, lobular, medullary, papillary, colloid (mucinous), or tubular histologies are allowed
3. Any receptor status is allowed (ER/PR/Her2-neu)
4. Patients with negative resection margins defined as 2 mm from ink, or a negative re-excision
5. Bilateral BC is allowed, provided each cancer meets inclusion criteria
6. Nodal RT is not allowed
7. There must be no concern for distant metastatic disease
8. Neoadjuvant or adjuvant chemotherapy is permitted provided pretreatment clinical and radiographic staging meets inclusion criteria. Specific adjuvant/neoadjuvant therapies are at the discretion of the treating Medical Oncologist. There are no systemic therapies that are not allowed on this study.
9. Patients must be deemed fit to receive the prescribed systemic therapy
10. Immunotherapy is allowed
11. Targeted Her-2 neu therapy, including concurrent therapy is allowed
12. Other targeted therapies are allowed (including but not limited to CDK inhibitors)
13. Endocrine therapy, including concurrent therapy is allowed
14. Participation in other non-RT clinical trial is allowed
15. Must be able to sign informed consent

Exclusion Criteria:

1. Patients with stage IV BC
2. Surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation. (If surgical margins are rendered free of disease by re-excision, the patient is eligible)
3. Prior thoracic or breast RT
4. The following RT methods and techniques are not permitted:

   * Brachytherapy or intraoperative RT (IORT)
   * Proton therapy
   * Regional nodal RT
   * Tumor bed boost
5. Patients who have breast reconstruction with implant or expander
6. Patients who have had a mastectomy for current BC
7. Patients requiring a tumor bed boost
8. Palpable or radiographic suspicious or contralateral lymph nodes or N2 disease
9. Paget's disease of the nipple.
10. Non-epithelial breast malignancies such as sarcoma or lymphoma
11. History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior to study entry
12. Active collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma
13. Pregnancy or lactation at the time of study entry/ or intention to become pregnant during treatment.
14. Patients with serious medical illness or psychiatric illness that would interfere with the trial.
15. Patients with active infection in the radiation treatment portal.

Ages: 60 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary(1) | up to 3 months
  Incidence of acute toxicities during and up to 3 months following completion of RT in BC patients who receive ultrahypofractionated WBI in BC patients who have received prior chemotherapy compared to historic controls for BC patients who have received prior chemotherapy and hypofractionated RT
Primary (2) | Up to 2 years
  Incidence of late toxicities of the breast up to 2 years following completion of RT in BC patients who receive ultrahypofractionated WBI in BC patients who have received prior chemotherapy compared to historic controls for BC patients who have received prior chemotherapy and hypofractionated RT

SECONDARY OUTCOMES:
Secondary (1) | Up to 3 months
  Incidence of acute toxicities during and up to 3 months following completion of RT for BC patients who received neoadjuvant chemotherapy vs adjuvant chemotherapy
Secondary (2) | Up to 2 years
  Incidence of late toxicities of the breast up to 2 years following completion of RT in BC patients who received neoadjuvant chemotherapy vs adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Russo, MD, Principal Investigator — MetroHealth Medical Center

IPD SHARING:
Plan to Share IPD: No